CLINICAL TRIAL: NCT07046247
Title: EFFECT OF TEFLON IMPLANT ON NERVE TISSUE AND ITS RELATIONSHIP WITH RECURRENCES IN THE TREATMENT OF TRIGEMINAL NEURALGIA BY MICROVASCULAR DECOMPRESSION, WITH SPECIAL ATTENTION TO THE METHOD OF APPLICATION. A RETROSPECTIVE CLINICAL STUDY.
Brief Title: Impact of Teflon Implantation Technique on Nervous Tissue and Recurrence Rates Following Microvascular Decompression for Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Vicente Vanaclocha, University Professor, University of Valencia
Other Study IDs: 188/2020
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Trigeminal Neuralgia; Microvascular Decompression; Teflon
Keywords: Trigeminal Neuralgia; Microvascular Decompression; Teflon Implant; Neurosurgical Techniques; Postoperative Complications; Magnetic Resonance Imaging
MeSH Terms: conditions — Trigeminal Neuralgia; Postoperative Complications | interventions — Microvascular Decompression Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Teflon pledgets group: Is the group of patients submitted to microvascular decompression for trigeminal neuralgia in whom the material to separate the trigeminal nerve from the offending vessel will be Teflon, placed in the form of one or more pledgets between the nerve and the vessel.
  Interventions: Procedure: Microvascular decompression for trigeminal neuralgia
- Shredded Teflon group: Is the group of patients submitted to microvascular decompression for trigeminal neuralgia in whom the material to separate the trigeminal nerve from the offending vessel will be shredded Teflon, placed around the displaced vessel away from the trigeminal nerve, aiming to induce a localized arachnoiditis away from the nerve that will fix the vessel in its new position, without any contact between the nerve and the vessel or the Teflon implant.
  Interventions: Procedure: Microvascular decompression for trigeminal neuralgia

INTERVENTIONS:
Procedure: Microvascular decompression for trigeminal neuralgia — Microvascular decompression for trigeminal neuralgia comparing two different forms to apply the Teflon implant

SUMMARY:
The study aims to see if shredded Teflon placed away from the trigeminal nerve is equally effective in pain control in Trigeminal Neuralgia while minimizing the risks of pain recurrence due to granuloma formation when this material is placed immediately close to the nerve in a pledget form.

DETAILED DESCRIPTION:
Complications associated with Teflon implants in the treatment of Trigeminal Neuraglia have been reported, including granuloma formation and persistent neuroinflammation, which can mimic tumor recurrence or lead to renewed symptoms. These concerns underscore the importance of precise implant positioning and accurate volume control. In our institution, we have consistently used a technique involving minimal amounts of shredded Teflon placed around the offending vessel, far from the trigeminal nerve itself. The goal is to elicit localized arachnoiditis to stabilize the artery and prevent re-compression. To our knowledge, to date, there are no published studies directly correlating the amount and form of Teflon used with subsequent inflammation and recurrence, particularly with imaging-based validation. Our study aims to fill this gap by retrospectively analyzing the outcomes of MVD procedures performed using this specific Teflon application method, correlating clinical outcomes with MRI findings to assess the degree of inflammatory response and the likelihood of symptom recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Trigeminal Neuralgia refractory to medical therapy and treated via microvascular decompression

Exclusion Criteria:

* Other craniofacial neuralgias, atypical facial pain, trigeminal neuralgia (TN) due to non-vascular causes (e.g., multiple sclerosis), and those with posterior fossa pathology, such as tumors, infarctions, hematomas, infections, or inflammatory lesions
* Patients treated by alternative methods, including percutaneous radiofrequency thermocoagulation, glycerol injection, balloon compression, or radiosurgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Trigeminal Neuralgia treated with microvascular decompression
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Modified Ranking scale | 5 years
  The Modified Rankin Scale (mRS) will be used to evaluate neurological disability, ranging from 0 (no symptoms) to 6 (death)
Barrow Neurological Institute Pain Intensity Scale | 5 years
  The Barrow Neurological Institute (BNI) Pain Intensity Scale will be used to assess pain control, ranging from 1 (no pain, no medication) to 5 (severe pain without relief)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Moratal, Secretary, Study Director — Fundación Consorcio Hospital General Universitario de Valencia
Locations (1):
- Consorcio Hospital General Universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Once the study is finised we will decide what to do

REFERENCES:
- [Background] Sindou M, Leston J, Decullier E, Chapuis F. Microvascular decompression for primary trigeminal neuralgia: long-term effectiveness and prognostic factors in a series of 362 consecutive patients with clear-cut neurovascular conflicts who underwent pure decompression. J Neurosurg. 2007 Dec;107(6):1144-53. doi: 10.3171/JNS-07/12/1144. PMID 18077952
- [Background] Pressman E, Jha RT, Zavadskiy G, Kumar JI, van Loveren H, van Gompel JJ, Agazzi S. Teflon or Ivalon(R): a scoping review of implants used in microvascular decompression for trigeminal neuralgia. Neurosurg Rev. 2020 Feb;43(1):79-86. doi: 10.1007/s10143-019-01187-0. Epub 2019 Nov 30. PMID 31786660
- [Background] Capelle HH, Brandis A, Tschan CA, Krauss JK. Treatment of recurrent trigeminal neuralgia due to Teflon granuloma. J Headache Pain. 2010 Aug;11(4):339-44. doi: 10.1007/s10194-010-0213-4. Epub 2010 Apr 24. PMID 20419329
- [Background] Deep NL, Graffeo CS, Copeland WR 3rd, Link MJ, Atkinson JL, Neff BA, Raghunathan A, Carlson ML. Teflon granulomas mimicking cerebellopontine angle tumors following microvascular decompression. Laryngoscope. 2017 Mar;127(3):715-719. doi: 10.1002/lary.26126. Epub 2016 Jun 19. PMID 27320780
- [Background] Prasetya M, Adidharma P, Inoue T, Sulistyanto A, Fadhil, Oswari S, Keswani RR, Kusdiansah M, Aji YK, Arham A. Case report: Teflon granuloma following microvascular decompression manifesting as light-triggered trigeminal neuralgia. Front Surg. 2022 Jul 22;9:904434. doi: 10.3389/fsurg.2022.904434. eCollection 2022. PMID 36570809
- [Background] Sindou M, Leston JM, Decullier E, Chapuis F. Microvascular decompression for trigeminal neuralgia: the importance of a noncompressive technique--Kaplan-Meier analysis in a consecutive series of 330 patients. Neurosurgery. 2008 Oct;63(4 Suppl 2):341-50; discussion 350-1. doi: 10.1227/01.NEU.0000327022.79171.D6. PMID 18981841
- [Background] Zheng JH, Sun K, Zhang HT, Xie YJ, Wang-Yang LX, Chen HY, Wang C. A Study on the Recurrence Rate of Trigeminal Neuralgia after MVD and the Related Factors. J Neurol Surg B Skull Base. 2020 Oct;81(5):572-578. doi: 10.1055/s-0039-1692687. Epub 2019 Jul 24. PMID 33134025
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Background] Okon II, Menon SS, Osama M, Aiman M, Paleare LFF, Eliseo DL 3rd, Shafqat MD, Ezeaku CO, Ferreira MY, Razouqi Y, Kapsetaki M, Saniel JDR, Panit NM, Rao AG, Iqbal U, Otobo DD, Alkhawaldeh IM, Pereira FS, Akbar I, Kasimieh O, Chaurasia B. Microvascular decompression: a contemporary update. BMC Surg. 2025 Jan 11;25(1):20. doi: 10.1186/s12893-025-02762-7. PMID 39794712
- [Background] Amaya Pascasio L, De La Casa-Fages B, Esteban de Antonio E, Grandas F, Garcia-Leal R, Ruiz Juretschke F. Microvascular decompression for trigeminal neuralgia: A retrospective analysis of long-term outcomes and prognostic factors. Neurologia (Engl Ed). 2021 May 25:S0213-4853(21)00071-2. doi: 10.1016/j.nrl.2021.03.009. Online ahead of print. English, Spanish. PMID 34049739